CLINICAL TRIAL: NCT00223613
Title: Intranasal Insulin for Prevention of Type 1 Diabetes in Children Carrying Increased HLA-Conferred Genetic Risk
Brief Title: Intranasal Insulin for Prevention of Type 1 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turku (Other)
Collaborators: Oulu University Hospital (Other); Tampere University (Other); University of Helsinki (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DIPP19942014; JDRF File # 4-1999-731
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2005-08

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; juvenile diabetes; insulin deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

INTERVENTIONS:
Drug: daily intranasal administration of insulin

SUMMARY:
Children born in Turku, Oulu and Tampere university cities in Finland are screened at birth for HLA alleles that carry increased risk to or protection from development of type 1 diabetes. Children carrying increased risk are followed at 3-12-month intervals for development of diabetes-associated autoantibodies. Children having at least two types of autoantibodies (of the four measured) in at least two consecutively drawn samples are randomized to receive daily intranasal insulin or placebo in a double-blinded 1:1 trial. Hypothesis is that intranasal insulin delays or prevents development of clinical type 1 diabetes. The primary outcome measure is development of clinical diabetes.

DETAILED DESCRIPTION:
Children born in Turku, Oulu and Tampere university cities in Finland are screened at birth for the HLA-DQB1 and DQA1 alleles that carry increased risk to or protection from development of type 1 diabetes. Children carrying increased risk are followed at 3-month intervals until 2 years of age and then at 6-12-month intervals until,15 years of age for development of diabetes-associated autoantibodies (autoantibodies against islet cells, insulin, glutamic acid decarboxylase and IA-2 protein). Children having at least two types of autoantibodies of the four measured in at least two consecutively drawn samples are randomized to receive daily intranasal insulin or placebo in a double-blinded 1:1 trial. Hypothesis is that intranasal insulin delays or prevents development of clinical type 1 diabetes. The primary outcome measure is development of clinical diabetes, but serum concentrations of autoantibodies, responses to intravenous glucose tolerance test and possible side effects of therapy are also closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* children carrying HLA-conferred genetic risk for developing type 1 diabetes
* have had at least two types of autoantibodies of ICA, IAA, GADA and IA-2A in at least two consecutive blood samples drawn at least 3 months apart
* age at least one year

Exclusion Criteria:

* severe other disease
* age above 15 years

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240
Dates: Start 1997-08; Study Completion 2005-08

PRIMARY OUTCOMES:
Development of clinical type 1 diabetes

SECONDARY OUTCOMES:
Number and concentration in serum of diabetes-associated autoantibodies (ICA, IAA, GADA and IA-2A)
Responses to intravenous glucose tolerance test
Possible side effects of therapy including hypoglycemia
Changes in serum metabolite patterns (metabolomics)

CONTACTS AND LOCATIONS:
Overall Officials: Olli G Simell, MD, PhD, Principal Investigator — University of Turku, Turku, Finland
Locations (1):
- Department of Pediatrics, University of Turku, Turku, Finland

REFERENCES:
- [Background] Kupila A, Sipila J, Keskinen P, Simell T, Knip M, Pulkki K, Simell O. Intranasally administered insulin intended for prevention of type 1 diabetes--a safety study in healthy adults. Diabetes Metab Res Rev. 2003 Sep-Oct;19(5):415-20. doi: 10.1002/dmrr.397. PMID 12951650
- [Background] Keskinen P, Korhonen S, Kupila A, Veijola R, Erkkila S, Savolainen H, Arvilommi P, Simell T, Ilonen J, Knip M, Simell O. First-phase insulin response in young healthy children at genetic and immunological risk for Type I diabetes. Diabetologia. 2002 Dec;45(12):1639-48. doi: 10.1007/s00125-002-0981-8. Epub 2002 Oct 30. PMID 12488953
- [Background] Kupila A, Keskinen P, Simell T, Erkkila S, Arvilommi P, Korhonen S, Kimpimaki T, Sjoroos M, Ronkainen M, Ilonen J, Knip M, Simell O. Genetic risk determines the emergence of diabetes-associated autoantibodies in young children. Diabetes. 2002 Mar;51(3):646-51. doi: 10.2337/diabetes.51.3.646. PMID 11872662
- [Background] Hermann R, Mantere J, Lipponen K, Veijola R, Soltesz G, Otonkoski T, Simell O, Knip M, Ilonen J. Lack of association of PAX4 gene with type 1 diabetes in the Finnish and Hungarian populations. Diabetes. 2005 Sep;54(9):2816-9. doi: 10.2337/diabetes.54.9.2816. PMID 16123375
- [Background] Kukko M, Toivonen A, Kupila A, Korhonen S, Keskinen P, Veijola R, Virtanen SM, Ilonen J, Simell O, Knip M. Familial clustering of beta-cell autoimmunity in initially non-diabetic children. Diabetes Metab Res Rev. 2006 Jan-Feb;22(1):53-8. doi: 10.1002/dmrr.584. PMID 16100734
- [Derived] Virtanen SM, Nevalainen J, Kronberg-Kippila C, Ahonen S, Tapanainen H, Uusitalo L, Takkinen HM, Niinisto S, Ovaskainen ML, Kenward MG, Veijola R, Ilonen J, Simell O, Knip M. Food consumption and advanced beta cell autoimmunity in young children with HLA-conferred susceptibility to type 1 diabetes: a nested case-control design. Am J Clin Nutr. 2012 Feb;95(2):471-8. doi: 10.3945/ajcn.111.018879. Epub 2012 Jan 11. PMID 22237062
- [Derived] Goldstein E, Hermann R, Renfors TJ, Nanto-Salonen KM, Korhonen T, Karkkainen M, Veijola RK, Knip M, Simell TT, Simell OG. From genetic risk awareness to overt type 1 diabetes: parental stress in a placebo-controlled prevention trial. Diabetes Care. 2009 Dec;32(12):2181-3. doi: 10.2337/dc09-0423. Epub 2009 Sep 14. PMID 19752173
- [Derived] Nanto-Salonen K, Kupila A, Simell S, Siljander H, Salonsaari T, Hekkala A, Korhonen S, Erkkola R, Sipila JI, Haavisto L, Siltala M, Tuominen J, Hakalax J, Hyoty H, Ilonen J, Veijola R, Simell T, Knip M, Simell O. Nasal insulin to prevent type 1 diabetes in children with HLA genotypes and autoantibodies conferring increased risk of disease: a double-blind, randomised controlled trial. Lancet. 2008 Nov 15;372(9651):1746-55. doi: 10.1016/S0140-6736(08)61309-4. Epub 2008 Sep 22. PMID 18814906